CLINICAL TRIAL: NCT02037230
Title: DOSE ESCALATION TRIAL OF THE Wee1 INHIBITOR AZD1775, IN COMBINATION WITH GEMCITABINE (+RADIATION) FOR PATIENTS WITH UNRESECTABLE ADENOCARCINOMA OF THE PANCREAS
Brief Title: Dose Escalation Trial of AZD1775 and Gemcitabine (+Radiation) for Unresectable Adenocarcinoma of the Pancreas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2013.094; HUM00079048 (Other: University of Michigan); NCT01916551 (obsolete NCT alias)
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Results first posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Adenocarcinoma of the Pancreas
MeSH Terms: interventions — adavosertib; Gemcitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MK-1775/ Gemcitabine/ Radiation Therapy (Experimental)
  Interventions: Drug: MK-1775; Drug: Gemcitabine; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: MK-1775 — MK-1775 will be given as an oral capsule on days 1 and 2, and on days 8 and 9 of every 3-week cycle .
Drug: Gemcitabine — Gemcitabine 1000mg/m2 will be infused over 30 minutes on days 1 and 8 of a 3 -week treatment cycle.
Radiation: Radiation Therapy — 52.5Gy in 25 fractions (2.1Gy/fraction), using intensity modulated radiation therapy (IMRT). Radiation therapy will be administered after chemotherapy.

SUMMARY:
The investigators' long-term goal is to improve the survival of patients with pancreatic cancer by enhancing the efficacy of gemcitabine-radiation by adding the Wee1 inhibitor MK-1775.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed adenocarcinoma of the pancreas.
* Patients will have unresectable disease, defined radiographically as >180 degrees involvement of the superior mesenteric artery or celiac trunk or SMV/portal vein impingement that cannot be surgically reconstructed, in the absence of distant metastasis..
* Patients must have a Zubrod performance status (measure of general well being that ranges from 0 to 5 where 0 represents perfect health) of < 2.
* Patients must have adequate organ function defined as follows: absolute neutrophil count of ≥ 1500/mm3, platelets ≥ 100,000/mm3, serum creatinine ≤ 2 mg/dl, total bilirubin ≤ 3, (with relief of biliary obstruction if present (PTC tube or endobiliary stent)) and AST < 5 times the upper limit of normal.
* Patients of reproductive potential must agree to use an effective contraceptive method during participation in this trial and for 6 months after the trial. Patients must not be breastfeeding.
* Patients must be aware of the investigational nature of the therapy and provide written informed consent.
* Patients must be at least 18 years old.

Exclusion Criteria:

* Other serious uncontrolled concomitant systemic disorders or psychiatric condition that would interfere with the safe delivery of protocol therapy.
* A history of previous chemotherapy for pancreatic cancer or abdominal radiation therapy.
* The use of any investigational agent in the month before enrollment into the study.
* Inability to discontinue a prescription or non-prescription drugs or other products known to be metabolized by CYP3A4, or to inhibit or induce CYP3A4 prior to Day 1 of dosing and to withhold throughout the study until 2 weeks after the last dose of study medication. Medications of particular concern are the following inhibitors of CYP3A4: azole antifungals (ketoconazole itraconazole, fluconazole and voriconazole), macrolide antibiotics (erythromycin, clarithromycin), cimetidine, aprepitant, HIV protease inhibitors, nefazodone and the following inducers of CYP3A4: phenytoin, barbiturates and rifampicin. Substrates of CYP3A4 include statins (lovastatin, simvastatin), midazolam, terfenadine, astemizole, and cisapride.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-01; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Lawrence, M.D., Ph.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Cuneo KC, Morgan MA, Sahai V, Schipper MJ, Parsels LA, Parsels JD, Devasia T, Al-Hawaray M, Cho CS, Nathan H, Maybaum J, Zalupski MM, Lawrence TS. Dose Escalation Trial of the Wee1 Inhibitor Adavosertib (AZD1775) in Combination With Gemcitabine and Radiation for Patients With Locally Advanced Pancreatic Cancer. J Clin Oncol. 2019 Oct 10;37(29):2643-2650. doi: 10.1200/JCO.19.00730. Epub 2019 Aug 9. PMID 31398082

RESULTS

PARTICIPANT FLOW:
Groups:
- AZD-1775 100 mg: AZD-1775 (MK-1775) 100 mg will be given as an oral capsule on days 1 and 2, and on days 8 and 9 of every 3-week cycle .
  Gemcitabine 1000mg/m2 will be infused over 30 minutes on days 1 and 8 of a 3 -week treatment cycle.
  Radiation Therapy: 52.5Gy in 25 fractions (2.1Gy/fraction), using intensity modulated radiation therapy (IMRT). Radiation therapy will be administered after chemotherapy. only in cycles 2 and 3
- AZD-1775 125 mg: AZD-1775 (MK-1775) 125 mg will be given as an oral capsule on days 1 and 2, and on days 8 and 9 of every 3-week cycle .
  Gemcitabine 1000mg/m2 will be infused over 30 minutes on days 1 and 8 of a 3 -week treatment cycle.
  Radiation Therapy: 52.5Gy in 25 fractions (2.1Gy/fraction), using intensity modulated radiation therapy (IMRT). Radiation therapy will be administered after chemotherapy. only in cycles 2 and 3
- AZD-1775 150 mg: AZD-1775 (MK-1775) 150 mg will be given as an oral capsule on days 1 and 2, and on days 8 and 9 of every 3-week cycle .
  Gemcitabine 1000mg/m2 will be infused over 30 minutes on days 1 and 8 of a 3 -week treatment cycle.
  Radiation Therapy: 52.5Gy in 25 fractions (2.1Gy/fraction), using intensity modulated radiation therapy (IMRT). Radiation therapy will be administered after chemotherapy. only in cycles 2 and 3
- AZD-1775 175 mg: AZD-1775 (MK-1775) 175 mg will be given as an oral capsule on days 1 and 2, and on days 8 and 9 of every 3-week cycle .
  Gemcitabine 1000mg/m2 will be infused over 30 minutes on days 1 and 8 of a 3 -week treatment cycle.
  Radiation Therapy: 52.5Gy in 25 fractions (2.1Gy/fraction), using intensity modulated radiation therapy (IMRT). Radiation therapy will be administered after chemotherapy. only in cycles 2 and 3
Period: Overall Study
Arm/Group | AZD-1775 100 mg | AZD-1775 125 mg | AZD-1775 150 mg | AZD-1775 175 mg
Started | 1 | 13 | 9 | 11
Completed 4 Cycles of Treatment | 1 | 9 | 7 | 9
Completed (Completed is defined as finishing 8 cycles of treatment) | 0 | 7 | 3 | 5
Not Completed | 1 | 6 | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD-1775 100 mg | AZD-1775 125 mg | AZD-1775 150 mg | AZD-1775 175 mg | Total
Number analyzed (Participants) | 1 | 13 | 9 | 11 | 34
Age, Continuous [Median (Full Range); unit: years] | 74 | 66 [54 to 78] | 62 [44 to 74] | 60 [52 to 73] | 68 [44 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 4 | 4 | 15
  Male | 0 | 7 | 5 | 7 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 1 | 11 | 9 | 10 | 31
  Unknown or Not Reported | 0 | 2 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 0 | 2
  White | 1 | 13 | 7 | 11 | 32
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of AZD1775 (MK-1775) When Used Concurrently With Gemcitabine and Radiation Therapy.
Description: Probability of dose limiting toxicities was calculated for each dose (p[DLT/d]) using the Time to Event Continual Reassessment Method (TITE-CRM). The target DLT rate was 0.30. Dose level 1 (150 mg AZD1775) was determined to be the MTD and recommended phase 2 dose (RP2D).
Time Frame: The observation period for MTD is defined as the first 4 cycles of treatment (with a 3 week break between cycle 3 and cycle 4), for a total of 105 days in length.
Population: All participants who received at least one dose of the study drug were evaluable for MTD.
Measure: Number; unit: mg
Groups:
- AZD1775 (MK-1775), Gemcitabine, Radiation Therapy: AZD1775 (MK-1775) will be given as an oral capsule on days 1 and 2, and on days 8 and 9 of every 3-week cycle .
  Gemcitabine 1000mg/m2 will be infused over 30 minutes on days 1 and 8 of a 3 -week treatment cycle.
  Radiation Therapy: 52.5Gy in 25 fractions (2.1Gy/fraction), using intensity modulated radiation therapy (IMRT). Radiation therapy will be administered after chemotherapy.
Arm/Group | AZD1775 (MK-1775), Gemcitabine, Radiation Therapy
Number analyzed (Participants) | 34
mg | 150

2. Secondary Outcome: Number of Patients With Phosphorylation Inhibition of Greater Than 0
Description: During the first cycle of treatment, patients underwent 2 biopsies: 3 h after treatment with gemcitabine (but before MK- 1775), and 2 hours after MK-1775. WEE1 signaling was assessed using immunohistochemistry (IHC) to measure phosphorylation of various markers including Cdk1 (Y15). Inhibition was quantified as the within subject change in the above markers between the two biopsy timepoints. Descriptive statistics of inhibition across subjects (for each marker) were calculated and reported by dose level.
Time Frame: First cycle of treatment
Population: 20 participants were evaluable for this outcome measure. Two sequential skin punch biopsies were obtained from 20 of the 34 study participants.
Measure: Number; unit: participants
Arm/Group | AZD-1775 100 mg | AZD-1775 125 mg | AZD-1775 150 mg | AZD-1775 175 mg
Number analyzed (Participants) | 1 | 8 | 5 | 6
participants | 1 | 7 | 3 | 5

3. Secondary Outcome: Overall Survival
Description: Overall survival (OS) summarized by Kaplan-Meier curves and characterized by descriptive statistics such as median OS. The time frame for data collection for OS varied depending on the length of patient follow-up, which ranged from 1.8 months to 47.2 months. Patients who enrolled soon after the study opened may have been followed longer than patients who enrolled later, toward the end of the study.
Time Frame: Up to 48 months following treatment
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | AZD-1775 100 mg | AZD-1775 125 mg | AZD-1775 150 mg | AZD-1775 175 mg
Number analyzed (Participants) | 1 | 13 | 9 | 11
months | 21.96 | 21.73 [16.67 to 39.81] | 23.84 [8.28 to 34.88] | 22.45 [6.81 to 25.35]

4. Secondary Outcome: Time From Date of Registration to Date of Documented Disease Progression
Description: Time from date of registration to date of documented disease progression summarized by Kaplan-Meier method. The time frame for data collection varied depending on the length of patient follow-up, which ranged from 1.8 months to 47.2 months. Patients who enrolled soon after the study opened may have been followed longer than patients who enrolled later, toward the end of the study.
Time Frame: Up to 48 months following treatment
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | AZD-1775 100 mg | AZD-1775 125 mg | AZD-1775 150 mg | AZD-1775 175 mg
Number analyzed (Participants) | 1 | 13 | 9 | 11
months | 8.05 | 9.44 [7.96 to 9.93] | 9.90 [4.90 to 18.02] | 6.08 [5.49 to 20.09]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the course of treatment (26 weeks). The time frame for data collection for all-cause mortality varied depending on the length of patient follow-up, which ranged from 1.8 months to 47.2 months. All-cause mortality includes all observed deaths while the study was ongoing, regardless of duration of patient follow-up. Patients who enrolled soon after the study opened may have been followed longer than patients who enrolled later, toward the end of the study.
Arm/Group | AZD-1775 100 mg | AZD-1775 125 mg | AZD-1775 150 mg | AZD-1775 175 mg
All-Cause Mortality (participants affected / at risk) | 1/1 | 9/13 | 5/9 | 6/11
Serious Adverse Events (participants affected / at risk) | 1/1 | 5/13 | 4/9 | 8/11
Other Adverse Events (participants affected / at risk) | 0/1 | 3/13 | 3/9 | 4/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD-1775 100 mg (N=1) | AZD-1775 125 mg (N=13) | AZD-1775 150 mg (N=9) | AZD-1775 175 mg (N=11)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ALT/AST elevation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anorexia, nausea/vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cholangitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GI bleed (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Septic shock (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolus (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Fever (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Altered mental status (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD-1775 100 mg (N=1) | AZD-1775 125 mg (N=13) | AZD-1775 150 mg (N=9) | AZD-1775 175 mg (N=11)
Pruritic Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Edema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-07): https://cdn.clinicaltrials.gov/large-docs/30/NCT02037230/Prot_SAP_000.pdf